CLINICAL TRIAL: NCT07277621
Title: Perceptions and Targeted Behavioral Change Interventions for Social Networking Site Addiction in School-going Adolescents of Karachi: A Concurrent Embedded Mixed-methods Case Study
Brief Title: Behavioral Interventions to Reduce Social Media Addiction Among School-Going Adolescents in Karachi
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Zaeema Ahmer, PhD Scholar, Dow University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-3760
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Internet Addiction Disorder
Keywords: Social media addiction; Behavioral change interventions
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): Description and content:
  Students in the intervention arm will receive a structured package of online, pre-recorded behavioral change videos specifically tailored for adolescents. Content domains include:
  Emotional regulation and coping skills
  Time management and self-monitoring of SNS use
  Sleep hygiene and evening routines
  Alternatives to SNS (physical activity, hobbies, face-to-face socializing)
  Awareness of risks, privacy, and cyber-safety
  Videos are short (5-8 minutes each), modular, and age-appropriate. The full intervention comprises 4 weekly modules delivered over 4 weeks, with follow-up reinforcement messages during weeks 5-12.
  Timing: Intervention delivered over 4 weeks, with follow-up assessments at 3 months post-baseline.
  Interventions: Behavioral: awareness videos
- control group (No Intervention): Description:
  Students in control schools will not receive the behavioral video intervention during the 3-month study period and will continue their usual school activities.
  Control group students will receive standard health promotion pamphlets unrelated to SNS behavior (to maintain basic equity of information) if required by school administration.
  After completion of follow-up data collection (3 months), the intervention package will be offered to control group students (delayed-intervention / wait-list) to ensure ethical fairness and benefit sharing.
  Timing: No active intervention during the 3-month evaluation window. Post-study access to intervention materials will be provided.

INTERVENTIONS:
Behavioral: awareness videos — this is a public health study whereby awareness videos will be shared with the intervention group to study behavior change for their addiction
  Arms: intervention arm

SUMMARY:
Addiction to Social Networking Sites (SNS) is considered a major public health problem and is well recognized around the world with serious social and health-related implications. There have been numerous studies that have been undertaken to examine the prevalence and severity of SNS addiction in Pakistani undergraduates. However, there are limited studies that have been done on the school-going adolescent population, especially in Pakistan. More importantly, there have been no interventions done to improve the minimization of the level of SNS addiction in this vulnerable cohort. This study will evaluate the effect of implementing targeted interventions for reducing the burden of SNS addiction so that in the future, evidence-based decisions may be taken and changes are incorporated in school curriculums.

Objective The specific objectives of this study are to estimate the prevalence of SNS addiction and to explore the perceptions of school-going adolescents regarding SNS addiction in metropolitan Karachi, Pakistan. It will further aim to introduce well-designed, online, tailored behavioral change interventions amongst students found with a high burden for significantly decreasing the prevalence of SNS addiction and for assessing their readiness to change.

Methodology This will be a mixed-methods concurrent embedded interventional study. The study will be conducted in selected private schools of Karachi in all its seven Districts. Prevalence will be assessed online by sharing an internationally validated tool with the students after getting students and their parent's consent. Concurrently, focus group discussions will be conducted in school premises with selected students from grades VI-XI. Once prevalence is ascertained, interventions will be designed to reduce levels of SNS addiction. Students will be randomly assigned to control and intervention groups and will be shown carefully designed interventions in the form of videos targeting specific domains of addiction. The effects of these interventions and readiness to change will be assessed after a period of three months.

DETAILED DESCRIPTION:
Addiction to Social Networking Sites (SNS) has emerged as a growing public health concern globally, with documented associations with psychological distress, academic decline, sleep disturbances, and impaired social functioning. While several studies in Pakistan have examined the prevalence and severity of SNS addiction among university students, there is a significant research gap concerning school-going adolescents-a population particularly vulnerable due to early and widespread digital exposure. Notably, no behavioral intervention studies have been conducted in Pakistan targeting the reduction of SNS addiction among adolescents. Addressing this gap is critical for informing preventive strategies and school-based digital wellness programs.

This study aims to assess the burden of SNS addiction among adolescents enrolled in private schools in Karachi and to evaluate the effectiveness of structured, online, behavioral change interventions tailored specifically for this age group. By generating actionable evidence, the study seeks to support future policy recommendations and integration of digital well-being content into school curricula.

Objectives

The primary objectives of this study are:

To estimate the prevalence and severity of Social Networking Site addiction among school-going adolescents in Karachi using an internationally validated assessment tool.

To explore perceptions, attitudes, and contextual factors influencing SNS overuse through focus group discussions with adolescents.

To implement and evaluate targeted behavioral change interventions, tailored to students identified with high levels of SNS addiction.

To assess readiness to change and the effect of the intervention on reducing SNS addiction scores over a three-month period.

Study Design

This research will employ a mixed-methods, concurrent embedded, quasi-experimental interventional design. Quantitative and qualitative components will be conducted simultaneously, with the quantitative arm functioning as the primary driver of the study and qualitative insights embedded to contextualize findings.

Study Setting

The study will be conducted in selected private schools across all seven districts of Karachi, Pakistan. Schools will be approached through administrative approval, and written consent/assent will be obtained from both parents and students as per ethical guidelines.

Study Procedures

1. Baseline Assessment

   An online, self-administered survey will be distributed to students (Grades VI-XI).

   The survey will include:

   Bergen Social Media Addiction Scale (BSMAS) & Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES), that are both internationally validated tools will be employed. Demographic information and patterns of SNS use will also be assessed.

   Students identified with moderate to high SNS addiction scores will qualify for the intervention phase.
2. Qualitative Component

Focus Group Discussions (FGDs) will be conducted with selected students to explore:

Perceptions about social media use

Motivations and triggers for excessive use

Barriers to reducing screen time

Suggestions for acceptable intervention formats

FGDs will be conducted on school premises by trained facilitators.

Intervention Phase

Eligible students will be assigned to Intervention or Control groups based on school logistics and administrative feasibility (non-random assignment).

The intervention group will receive online, pre-recorded, culturally tailored behavioral change videos addressing:

Digital hygiene and time management

Emotional regulation

Sleep hygiene

Healthy alternative activities

Risks of excessive social media use

The control group will continue usual routines and will be offered the intervention later.

4. Follow-up and Outcome Assessment

After three months, both groups will complete the BSMAS & SOCRATES again.

Primary Outcome: Change in SNS addiction scores from baseline to three months.

Secondary Outcomes:

Self-reported changes in screen time

Improvement in readiness to change (using adapted readiness-to-change scales)

Sample Size

A sample size of approximately 260 students (130 per group) is planned, accounting for anticipated attrition.

Significance of the Study

This will be the first interventional study in Pakistan evaluating structured behavioral strategies to reduce SNS addiction among adolescents. The results will provide critical evidence to support:

Integration of digital wellness modules into school curricula

Development of adolescent-centered mental health promotion strategies

Early preventive interventions for problematic technology use

By adopting a mixed-methods approach, the study will not only quantify addiction levels but also explore contextual influences, making the findings more relevant for policy, program design, and future research.

ELIGIBILITY:
Inclusion Criteria:

* Age between 11-16 years
* Either male or female (or any other gender)
* User of any of the listed social media (Facebook, Instagram, WhatsApp, YouTube, Snapchat, Tumblr, TikTok or Discord) for the past one year
* In possession of a functioning laptop/smartphone for attending online intervention vlogs and receiving text messages

Exclusion Criteria:

* Any student undergoing psychiatric or psychological treatment/ counseling
* Any student taking anti-psychotics or any treatment for chronic disorders (diabetes, cancer, kidney disease, asthma)
* Any student suffering from chronic mental illness, e.g. depression, anxiety, schizophrenia, etc.
* Any student who has suffered a major trauma in the past year, e.g. death of a loved one, accident, etc.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in Social Networking Site Addiction Score using Bergen Social Media Addiction Scale (BSMAS) | from baseline to 3 months post intervention
  This outcome will assess the change in social networking site addiction levels among participating adolescents from baseline to 3 months follow-up. The Bergen Social Media Addiction Scale (BSMAS), a validated 6-item self-report tool, will be used to measure addiction severity. Each item is scored on a 5-point Likert scale (1-5), yielding a total score range of 6 to 30, with higher scores indicating greater risk of addiction.
  Unit of Measure:
  Score (range 6-30) (Change in total BSMAS score from baseline to 3-month follow-up)
Readiness to Change Score using the Readiness to Change Questionnaire (SOCRATES - Adapted for SNS use) | intervention for a month and follow-up of 3 months
  Readiness to change problematic social networking site (SNS) use will be assessed using the SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) adapted specifically for SNS behaviors.
  The SOCRATES tool consists of three subscales:
  Recognition - awareness of problematic SNS use
  Ambivalence - uncertainty about behavior change
  Taking Steps - active efforts to reduce problematic SNS use
  Participants respond to Likert-scale items (1-5), and subscale scores are summed to generate total scores for each domain. Higher scores indicate greater readiness and motivation to change SNS-related behaviors.
  Unit of Measure:
  Subscale Score (continuous)
  Recognition Score (range depends on adapted item count)
  Ambivalence Score
  Taking Steps Score

CONTACTS AND LOCATIONS:
Overall Officials: Zaeema Ahmer, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of health Sciences, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the present study are not publicly available. However, they are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Requests should be made to corresponding author for access